CLINICAL TRIAL: NCT02269007
Title: A Phase I Clinical Trial for Inactivated Quadrivalent Influenza Vaccine (Split Virion) in Healthy Adults in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Jiangsu Jindike Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JSVCT019
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Influenza
Keywords: safety, tolerance, quadrivalent influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.5ml influenza vaccine (Experimental): 0.5ml inactivated quadrivalent influenza vaccine (split virion) for each subject, one dose
  Interventions: Biological: inactivated quadrivalent influenza vaccine (split virion)

INTERVENTIONS:
Biological: inactivated quadrivalent influenza vaccine (split virion) — 0.5ml inactivated quadrivalent influenza vaccine (split virion) for each subject, one dose

SUMMARY:
Influenza is an acute respiratory disease caused by influenza viruses. There are three types of the virus including A, B and C. Both type A and type B viruses can cause acute febrile respiratory tract infection, characterized by sudden fever, headache, muscle pain, cough, sore throat, nasal congestion and general malaise.

Influenza can periodically cause worldwide pandemic. For nearly a century, the influenza virus had occurred four large variation, causing three world pandemic. Studies have shown that since 1957, most of those new variants of influenza virus started in China, which is recognized by the world to have high incidence of influenza. At present, trivalent influenza vaccines are widely used in China. They only contain two kinds of type A virus antigens and one type B virus antigen. But since 2000, two kinds of type B strains (Victoria and Yamagata) have caused an alternating cycle in different seasons. Gradually, evolved from the original single lineage of influenza B virus B/Yamagata, two distinct antigenic lineages-B/Victoria and B/Yamagata have alternately dominated or caused a mix of popular lineage. These two lineages have little or nearly no cross-protection. Therefore, trivalent influenza vaccines may not cover the popular strains of influenza B virus, whereas quadrivalent influenza vaccines will help to simultaneously prevent two kinds of type A viruses and two kinds of type B virus.

DETAILED DESCRIPTION:
Influenza is an acute respiratory disease caused by influenza viruses. There are three types of the virus including A, B and C. Both type A and type B viruses can cause acute febrile respiratory tract infection, characterized by sudden fever, headache, muscle pain, cough, sore throat, nasal congestion and general malaise. The main transmission of influenza is through those highly contagious aerosol droplets containing influenza virus passed from infected people to susceptible population. Each year in the fall and winter infection of influenza is widespread in various age groups, with high incidence rate. Although influenza is generally a self-limiting disease, but in children, the elderly (especially those above 65 years old and those with chronic heart, lung, kidney, liver, blood or metabolic diseases such as diabetes or other certain diseases) and those with poor immunity function, influenza can easily lead to serious flu complications such as pneumonia, resulting in severe increase of morbidity and mortality.

Influenza can periodically cause worldwide pandemic. For nearly a century, the influenza virus had occurred four large variation, causing three world pandemic. Studies have shown that since 1957, most of those new variants of influenza virus started in China, which is recognized by the world to have high incidence of influenza. At present, trivalent influenza vaccines are widely used in China. They only contain two kinds of type A virus antigens and one type B virus antigen. But since 2000, two kinds of type B strains (Victoria and Yamagata) have caused an alternating cycle in different seasons. Gradually, evolved from the original single lineage of influenza B virus B/Yamagata, two distinct antigenic lineages-B/Victoria and B/Yamagata have alternately dominated or caused a mix of popular lineage. These two lineages have little or nearly no cross-protection. Therefore, trivalent influenza vaccines may not cover the popular strains of influenza B virus, whereas quadrivalent influenza vaccines will help to simultaneously prevent two kinds of type A viruses and two kinds of type B virus.

In order to evaluate safety and tolerance of the quadrivalent influenza vaccine produced by Jiangsu Jindike Biotechnology Co., Ltd. a phase I clinical trial is planned to conduct in healthy adults aged from 18 to 49 years in China.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 49 years old
* Healthy adults judged from medical history and clinical examination
* Subjects able to understand and sign the informed consent
* Subjects who can and will comply with the requirements of the protocol
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria:

* Subject who has a medical or family history of any of the following: allergic history, seizure, epilepsy, brain or mental disease
* Any prior administration of influenza vaccine in last 6 month
* Subject who is allergic to any ingredient of the vaccine
* Female subject with a positive result after urine pregnancy test or during pregnancy or baby nursing period
* Subject with damaged or low immune function which has already been known
* Subject who had a seasonal influenza medical history in last 6 months
* Subject with acute febrile illness or infectious disease
* Major congenital defects or serious chronic illness, including perinatal brain damage
* Thrombocytopenia, blood coagulation disorder or bleeding difficulties with intramuscular injection
* Subject who has serious allergic history
* Subject with other medical history not suitable for vaccination such as fainting during injection or acupuncture treatment
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of other research medicine/vaccine in last 30 days
* Any prior administration of any attenuated live vaccine in last 30 days
* Any prior administration of subunit or inactivated vaccines in last 14 days, such as pneumococcal vaccine
* Any medical, psychological, social or other condition judged by investigator, that may interfere subject's compliance with the protocol or signature on informed consent

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
to evaluate incidence of solicited adverse reactions (including systemic and local adverse reactions) after vaccination | 0-7 days after vaccination
  to evaluate incidence of solicited adverse reactions (including systemic and local adverse reactions) within 0-7 days after vaccination

SECONDARY OUTCOMES:
to evaluate incidence of unsolicited adverse reactions (including systemic and local adverse reactions) after vaccination | 0-21 days after vaccination
  to evaluate incidence of unsolicited adverse reactions (including systemic and local adverse reactions) within 0-21 days after vaccination
to evaluate incidence of serious adverse event (SAE) after vaccination | 0-21 days after vaccination
  to evaluate incidence of serious adverse event (SAE) within 0-21 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Fengcai Zhu, Master, Principal Investigator — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Guanyun County Center for Disease Control and Prevention, Liangyungang, Jiangsu, China